CLINICAL TRIAL: NCT05490160
Title: Alteration of Thrombelastography and Hemostatic Function in Patients Undergoing Total Knee Arthroplasty With Intra-articular Tranexamic Acid Administration
Brief Title: Alteration of Thrombelastography and Coagulation Function in Patients Undergoing Total Knee Arthroplasty With Intra-articular Tranexamic Acid Administration
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IIT-2022-0059
Record Dates: First submitted 2022-08-01; First posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-07

CONDITIONS: Arthropathy of Knee
Keywords: Total Knee Arthroplasty; Thrombelastography; Coagulation Function
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tranexamic acid group: During the total knee arthroplasty, the patients received a 2-g retrograde injection of tranexamic acid through the drain after closure, with subsequent clamping of the drain for 6 hours.
  Interventions: Drug: Tranexamic acid
- Non-tranexamic acid group: During the total knee arthroplasty, the patients did not receive tranexamic acid administration.

INTERVENTIONS:
Drug: Tranexamic acid — During the total knee arthroplasty, the patients received a 2-g retrograde injection of tranexamic acid through the drain after closure, with subsequent clamping of the drain for 6 hours.
  Groups: Tranexamic acid group

SUMMARY:
The main aim and scope of this study is making comparison about the thrombelastography and coagulation function in patients before and after the total knee arthroplasty with intra-articular tranexamic acid administration. The results may identify the influence of the intra-articular tranexamic acid administration on the relative coagulability monitoring.

ELIGIBILITY:
Inclusion Criteria:

* The patients received primary total knee arthroplasty;
* Normal pre-operative coagulation function;
* Complete surgery document, transfusion document and relative blood test.

Exclusion Criteria:

* The patients received complicated total knee arthroplasty;
* Abnormal pre-operative coagulation function caused by some diseases such as hepatic inadequacy, thrombocytopenia et al.
* Incomplete documents.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients received primary total knee arthroplasty.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2022-08-05 (Estimated); Primary Completion 2022-08-20 (Estimated); Study Completion 2022-08-28 (Estimated)

PRIMARY OUTCOMES:
R time | day0 (pre-operative)
  R time is the period from the initiation of the thrombelastography test till the beginning of the clot formation.
R time | day3 (post-operative)
  R time is the period from the initiation of the thrombelastography test till the beginning of the clot formation.
K time | day0 (pre-operative)
  K time is the period from the start of the clot formation to the curve reaches amplitude of 20mm in the thrombelastography.
K time | day3 (post-operative)
  K time is the period from the start of the clot formation to the curve reaches amplitude of 20mm in the thrombelastography.
Alpha angle | day0 (pre-operative)
  Alpha angle is the angle between the baseline and the tangent to the thrombelastography curve through the starting point of coagulation.
Alpha angle | day3 (post-operative)
  Alpha angle is the angle between the baseline and the tangent to the thrombelastography curve through the starting point of coagulation.
Maximal amplitude (MA) | day0 (pre-operative)
  Maximal amplitude (MA) is a direct measure of the highest point on the thrombelastography curve and represents clot strength.
Maximal amplitude (MA) | day3 (post-operative)
  Maximal amplitude (MA) is a direct measure of the highest point on the thrombelastography curve and represents clot strength.
Clot index (CI) | day0 (pre-operative)
  Clot index (CI) represents the haemostasis profile and is calculated based on R time, K time, Alpha angle and MA parameters.
Clot index (CI) | day3 (post-operative)
  Clot index (CI) represents the haemostasis profile and is calculated based on R time, K time, Alpha angle and MA parameters.

SECONDARY OUTCOMES:
Prothrombin time (PT) | day0 (pre-operative)
  Prothrombin time (PT) is one of the parameters which reflects the coagulation function.
Prothrombin time (PT) | day3 (post-operative)
  Prothrombin time (PT) is one of the parameters which reflects the coagulation function.
Activated partial thromboplastin time (APTT) | day0 (pre-operative)
  Activated partial thromboplastin time (APTT) is one of the parameters which reflects the coagulation function.
Activated partial thromboplastin time (APTT) | day3 (post-operative)
  Activated partial thromboplastin time (APTT) is one of the parameters which reflects the coagulation function.
Hemoglobin in g/L | day0 (pre-operative)
  Hemoglobin is a parameter which reflects the blood loss or anemia.
Hemoglobin in g/L | day3 (post-operative)
  Hemoglobin is a parameter which reflects the blood loss or anemia.
Red blood cell specific volume (HCT) | day0 (pre-operative)
  Red blood cell specific volume (HCT) is a parameter which reflects the ratio of the red blood cells in the whole blood.
Red blood cell specific volume (HCT) | day3 (post-operative)
  Red blood cell specific volume (HCT) is a parameter which reflects the ratio of the red blood cells in the whole blood.
Fibrinogen in g/L | day0 (pre-operative)
  Fibrinogen is one of the parameters which reflects the coagulation function.
Fibrinogen in g/L | day3 (post-operative)
  Fibrinogen is one of the parameters which reflects the coagulation function.
Platelet count in 10^9g/L | day0 (pre-operative)
  Plstelet count is a parameter which reflects the amount of the platelet in the whole blood.
Platelet count in 10^9g/L | day3 (post-operative)
  Plstelet count is a parameter which reflects the amount of the platelet in the whole blood.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Du, Study Chair — RenJi Hospital

IPD SHARING:
Plan to Share IPD: No